CLINICAL TRIAL: NCT06259409
Title: A Randomized Clinical Study Evaluating the Safety of Regenn® Negative Pressure Therapy System in Orthopaedic Surgical Wound Management
Brief Title: Regenn® Therapy System Safety Study
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Progenerative Medical, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Doc-0353
Record Dates: First submitted 2024-01-26; First posted 2024-02-14 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Surgical Wound
MeSH Terms: conditions — Surgical Wound | interventions — Negative-Pressure Wound Therapy

STUDY DESIGN:
Intervention Model Description: Prospective, randomized, controlled investigational study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Treatment Arm (Experimental): This group will receive the study device, Regenn® Negative Pressure Therapy System, a form of Negative Pressure Wound Therapy (NPWT). Regenn® Therapy manages the surgical wound by the application of reduced pressure therapy (i.e., mild vacuum). Reduced pressure therapy is controlled by a hand-sized, battery-operated pump and is delivered by an attached small, dressing that the surgeon places in the surgical wound at the end of the surgery. Reduced pressure therapy is applied while the patient recovers from surgery.
  Interventions: Device: Regenn® Negative Pressure Therapy System
- Control Arm (Active Comparator): This group will receive the control device, also a form of Negative Pressure Wound Therapy (NPWT), which manages the surgical wound by the application of reduced pressure therapy (i.e., mild vacuum). Reduced pressure therapy is controlled by a hand-sized, battery-operated pump and is delivered by a small tube connected to a wound dressing placed over the closed surgical wound at the end of the surgery. Reduced pressure therapy is applied while the patient recovers from surgery.
  Interventions: Device: Prevena™ Incision Management System

INTERVENTIONS:
Device: Regenn® Negative Pressure Therapy System — Controlled application of negative pressure (i.e., reduced atmospheric pressure or mild vacuum) to manage the wound environment.
  Other Names: NPWT; Negative Pressure Wound Therapy
  Arms: Treatment Arm
Device: Prevena™ Incision Management System — Controlled application of negative pressure (i.e., reduced atmospheric pressure or mild vacuum) to manage the wound environment.
  Other Names: NPWT; Negative Pressure Wound Therapy
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is to evaluate the safety of the investigational device, Regenn® Negative Pressure Therapy System (Regenn® Therapy), a form of Negative Pressure Wound Therapy (NPWT), in the post-operative surgical wounds of patients undergoing lumbar spinal fusion surgeries. The main questions the study aims to answer are:

* The device-related serious adverse event rate.
* Patient post-operative pain as assessed using a validated pain measurement scoring system.
* The number and type of adverse events.
* The rate of delayed seroma formation.

Participants will

* Be screened for their suitability to participate in the investigational study using questions about their health, medical history, and current medications.
* Undergo a physical exam, an assessment of patient vital signs and routine blood analyses.
* Complete an Informed Consent Form if selected to participate in the investigational study.
* Be randomly assigned to the different study arms.
* Not change the operation of their respective device or to disturb components of their device.
* Notify their surgeon or designated healthcare provider should they have any questions or encounter any issues with their device.
* Attend two post-operative visits at approximately one month and three months.

ELIGIBILITY:
Inclusion Criteria (must meet ALL):

* Subject has provided written informed consent on a form reviewed and approved by the Institutional Review Board for the clinical site.
* The subject is 18 - 80 years old.
* The subject has Spondylolisthesis of Meyerding Grade II or less, or has Degenerative Disc Disease (DDD) accompanied by back pain with or without leg pain at a level between L1 and S1 confirmed by history and radiographic assessment. DDD is determined to be present if one or more of the following are noted:

  * Instability (defined as angulation ≥ 5 degrees and/or translation ≥ 3mm on flexion/extension radiographs;
  * Osteophyte formation of facet joints or vertebral endplates;
  * Decreased disc height, on average by >2mm, but dependent upon the spinal level;
  * Scarring / thickening of ligamentum flavum, annulus fibrosis, or facet joint capsule;
  * Herniated nucleus pulposus;
  * Facet joint degeneration / changes; and/or
  * Vacuum phenomenon.
* Female subjects of childbearing potential must not be pregnant or nursing and must agree to use of contraception for the study duration. Female subjects who are surgically sterile or post-menopausal are exempt from having a pregnancy test and birth control.
* The subject is willing and able to comply with the protocol mandated follow-up visits and testing regimen.

Exclusion Criteria (candidates meeting ANY of the following at the time of the study procedure are NOT eligible):

* Subject is unable or unwilling to provide informed consent or is unable to conform to the study protocol follow-up procedures and visits.
* Subject has a contraindication (including allergic reaction) to antiplatelet/anticoagulant medications, nickel, titanium, bone allograft, or blood transfusion that is not amenable to pretreatment with steroids or/and antihistamines.
* Subject has a history of bleeding diatheses or coagulopathy.
* Subject has concomitant hepatic insufficiency, thrombophlebitis, uremia, systemic lupus erythematosus (SLE), or any autoimmune diseases.
* Subject is receiving dialysis or immunosuppressive therapy.
* Subject suffered a hemorrhagic stroke < 6 months prior to the study procedure.
* Subject is undergoing spinal surgery for vertebral fracture, trauma, or scoliosis.
* Subject has any form of active malignancy.
* Subject is an intravenous drug user and/or alcoholic.
* Subject is diagnosed with septicemia at the time of the study procedure.
* Subject is a smoker.
* Subject has Type I diabetes.
* Subject has overt, uncontrolled Type II diabetes.
* Subject has a condition requiring postoperative medications that would be expected to interfere with fusion (e.g., steroids), or has received drugs that interfere with bone metabolism within 2 weeks of the surgery.
* Subject is suffering from gross obesity, defined as > 40% IBW.
* Subject exhibits Waddell signs of Inorganic Behavior ≥ 3.
* Subject has had a previous, anterior spinal fusion, interbody spinal fusion, or posterior spinal instrumentation at the involved level.
* Subject has another medical condition, which may cause them to be non-compliant with the protocol, confound the data interpretation, or is associated with limited life expectancy of less than two years.
* Subject has a systemic disease of connective tissue such as Rheumatoid Arthritis, or Ankylosing Spondylitis.
* Subject is a prisoner.
* Subject is currently participating in an investigational drug or another device study that has not completed the primary endpoint or that clinically interferes with the study endpoints. (Note: Trials requiring extended follow-up for products that were investigational, but have since become commercially available, are not considered investigational trials).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Device-related Serious Adverse Event Rate | Post-operative follow ups at 2-8 weeks and 3-6 months.
  The device-related serious adverse event rate associated with the use of the investigational device and the comparator device. Wound complications requiring surgical intervention, such as wound dehiscence, will be the primary indicator of blood supply at the wound site, damage to the surrounding tissue, and progression of wound healing.

SECONDARY OUTCOMES:
Post-operative Pain Profile | Post-operative up to the 3-6 month follow up visit.
  Post-operative pain will be assessed using the Numerical Rating Scale (NRS), a validated pain measurement scoring system with a pain rating scale of 0 - 10, where zero means "No pain" and 10 means "The worst pain imaginable"
Adverse Events Related to the Investigational Device | Post-operative follow ups at approximately one month and three months.
  The number and type of adverse events associated with the use of the investigational device. Assessment will include wound complications not requiring surgical intervention, device complications, medical complications and infections complications.

OTHER OUTCOMES:
Delayed Seroma Formation Rate | Post-operative follow up at 2-8 weeks (at the surgeon's discretion) and at 3-6 months (required).
  Delayed seroma formation will be assessed by ultrasound imaging during post-operative follow up visits.

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Kansas Medical Center, Kansas City, Kansas, United States

IPD SHARING:
Plan to Share IPD: No